CLINICAL TRIAL: NCT05594524
Title: Body Confident Athletes: A Randomized Controlled Trial Testing the Efficacy of a Coach-Led Body Image Intervention for Adolescent Girls in Sport
Brief Title: Coach-Led Body Image Intervention for Girls in Sport - RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Unilever R&D (Industry); Nike (Industry); Tucker Center for Research on Girls & Women in Sport (University of Minnesota) (Unknown); Cairn Guidance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HAS.21.03.120c
Record Dates: First submitted 2022-10-12; First posted 2022-10-26 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Intervention; Waitlist Control
Keywords: Body image; Embodiment; Girls; Athletes; Coaches; Task shifting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Confident Athletes (Experimental): Participants in the intervention condition will take part in an in-person program consisting of three sessions over three weeks.
  Interventions: Behavioral: Body Confident Athletes
- Waitlist control (No Intervention): Participants will not be explicitly told their study condition, although they will be made aware of the assessment time points and whether they will receive access to the intervention after the first survey (intervention group) or after follow-up assessments (waitlist control group). Following completion of follow-up assessments, the control condition will get access to the intervention, but they will not be monitored or assessed.

INTERVENTIONS:
Behavioral: Body Confident Athletes — The Body Confident Athletes program is a three-session in-person program designed to be delivered by coaches to their athletes. Groups should be of approximately 10-20 girls. The sports organizations will work with the community partner and researchers on how to schedule the intervention over a three-week period. These sessions can replace a regular sport practice each week or an additional session can be organized by the sports organization. Each session will take approximately 60 minutes and will consist of four phases, including The Game Plan (5 mins), The Knowledge (20 mins), The Skills (20 mins), and The Final Score (15 mins). A variety of activity modalities will be utilized to convey learning outcomes, including group and individual activities and discussion-, writing-, and movement-based activities.
  Arms: Body Confident Athletes

SUMMARY:
According to the World Health Organization, only 15% of 11-17-year-old girls meet the recommended daily physical movement guidelines (e.g., 60 minutes per day). Despite extensive research highlighting the protective factors associated with sport on both mental and physical health, body image concerns are a key barrier to girls' participation in, and enjoyment of, sport. Sports-related environments and society more broadly further exacerbate these concerns through harmful gender stereotypes that perpetuate female objectification, discrimination, and harassment. This includes the promotion of unrealistic and sexualized appearances of female athletes, uncomfortable and objectifying uniforms, and appearance and competence-related teasing from male and female peers, as well as coaches.

The magnitude of this issue and how best to address it can be understood from a socioecological perspective. Researchers suggest developing multi-faceted and multi-tiered approaches that have scope for targeting the individual, interpersonal, organizational, and societal levels. The current research will test the first coach-led body image program for girls in sport. The Body Confident Athletes program was co-created with girls and coaches through an international multi-disciplinary partnership between academics, health professionals, industry, and community organizations. Multi-disciplinary partnerships can create a supportive landscape by upskilling girls and influential community members (e.g., coaches) in dealing with body image concerns, which will likely lead to sustained sports participation and biopsychosocial benefits.

As such, the aim of the present study is to conduct a large-scale randomized controlled trial (RCT) to evaluate the effectiveness of the Body Confident Athletes program. The program consists of three 60-minute sessions delivered by coaches to adolescent girls. Each session tackles a distinct theme related to body image in the sport context. Outcomes will be assessed at pre-intervention, post-intervention (three weeks later), and follow-up (at one and three months). Outcomes will include body image and sport enjoyment (primary outcomes); body appreciation, attuned self-care, resisting objectification, and positive and negative affect (secondary outcomes); and intervention acceptability, fidelity, and adherence (process outcomes). The comparison control arm will be a waitlist control condition.

To undertake this project, sports organizations will be cluster-randomized into the intervention group or the control group, with 800 girls anticipated in each arm. Those in the intervention condition will complete baseline assessments (target outcomes and demographic information), take part in the three-week intervention, and then complete the post-intervention and follow-up assessments (target and process outcomes). Those in the waitlist control condition will complete the baseline assessments (target outcomes and demographic information), a second assessment three weeks later (target outcomes only), and follow-up assessments after one and three months, after which they will get access to the intervention. However, their engagement with the intervention will not be monitored or assessed. At completion of the post-intervention survey, all participants will receive a debrief form, outlining the study aims and objectives, and support resources for body image and eating concerns.

The investigators hypothesize that girls who take part in the Body Confident Athletes intervention will report higher levels of body esteem, sport enjoyment, body appreciation, attuned self-care, resisting objectification, and positive affect and lower levels of negative affect at post-intervention and follow-up, compared to girls who do not take part in the intervention.

Note: This research has been approved by the University of the West of England Research Ethics Committee (ref no. HAS.21.03.120) and the University of Minnesota Institutional Review Board (ref no. STUDY00012457).

ELIGIBILITY:
Inclusion Criteria:

* Girls aged 11-17 years old
* English speaking
* Residing in the United States

Exclusion Criteria:

* n/a

Ages: 11 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — We will include girls in the current study, referring to the girl child defined as younger than 18 years old who was assigned female at birth and all individuals who identify as a girl.
Enrollment: 568 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-05-07 (Actual); Study Completion 2023-05-07 (Actual)

PRIMARY OUTCOMES:
Change in body esteem (assessed via the Body Esteem Scale for Adults and Adolescents) | Baseline, pre-intervention; immediately after the intervention (3 weeks later); 1 month after completion of the intervention; 3 months after completion of the intervention
  The Body Esteem Scale for Adults and Adolescents (BESAA) assesses body esteem (BE), which refers to self-evaluations of one's body or appearance. The BESAA has 3 subscales: BE-Appearance (general feelings about appearance), BE-Weight (weight satisfaction), and BE-Attribution (evaluations attributed to others about one's body and appearance). For the purposes of this study, only the BE-Appearance and BE-Weight subscales will be utilized. BESAA scores range from 0-4 with higher scores on the BESAA indicating higher levels of body esteem.
Change in sport enjoyment (assessed via the Sources of Enjoyment in Youth Sport Questionnaire) | Baseline, pre-intervention; immediately after the intervention (3 weeks later); 1 month after completion of the intervention; 3 months after completion of the intervention
  The Sources of Enjoyment in Youth Sport Questionnaire (SEYSQ) assesses the source of an athlete's enjoyment in sport according to two spectrums (intrinsic motivation vs. extrinsic motivation and achievement vs. non-achievement factors), resulting in four quadrants indicating the four sources of an athlete's enjoyment. SEYSQ scores range from 1-5.

SECONDARY OUTCOMES:
Change in body appreciation (assessed via the Body Appreciation Scale-2) | Baseline, pre-intervention; immediately after the intervention (3 weeks later); 1 month after completion of the intervention; 3 months after completion of the intervention
  The Body Appreciation Scale-2 (BAS-2) assesses body appreciation. Body appreciation has been associated positively with adaptive characteristics and negatively with maladaptive characteristics among samples of women and men from Western countries, including the United States, the United Kingdom, and Australia. BAS-2 scores range from 1-5 with higher scores on the BAS-2 indicating higher levels of body appreciation.
Change in attuned self-care (assessed via the Youth Experience of Embodiment Scale - Attuned Self-Care subscale) | Baseline, pre-intervention; immediately after the intervention (3 weeks later); 1 month after completion of the intervention; 3 months after completion of the intervention
  The Youth Experience of Embodiment Scale (YEES) assesses how girls inhabit their body (e.g., body connection and comfort, attuned self-care) and how they navigate the world (e.g., with agency, resisting self-objectification). Attuned self-care specifically reflects the degree of attunement and responsiveness to the embodied self and its physical, emotional, relational, aspirational, and spiritual needs. YEES scores range from 1-5 with higher scores on the YEES indicating higher levels of embodiment.
Change in resisting objectification (assessed via the Youth Experience of Embodiment Scale - Resisting Objectification subscale) | Baseline, pre-intervention; immediately after the intervention (3 weeks later); 1 month after completion of the intervention; 3 months after completion of the intervention
  The Youth Experience of Embodiment Scale (YEES) assesses how girls inhabit their body (e.g., body connection and comfort, attuned self-care) and how they navigate the world (e.g., with agency, resisting self-objectification). Resisting objectification specifically refers to inhabiting the body as a subjective site (vs. as an objectified site); i.e., the immersion in subjectively perceived embodied experiences and meaningful pursuits, and resistance to inhabiting the body as an object of gaze. YEES scores range from 1-5 with higher scores on the YEES indicating higher levels of embodiment.
Change in positive and negative affect (assessed via the 10-item Positive and Negative Affect Schedule for Children) | Baseline, pre-intervention; immediately after the intervention (3 weeks later); 1 month after completion of the intervention; 3 months after completion of the intervention
  The 10-item Positive and Negative Affect Schedule for Children (PANAS-C) is a self-report questionnaire that consists of two 5-item scales to measure positive and negative affect. Each item is rated on a 5-point scale of 1 (very slightly or not at all) to 5 (extremely). Higher levels on the positive and negative affect scales indicate higher levels of positive and negative affect, respectively.

OTHER OUTCOMES:
Total acceptability of the intervention (assessed via a self-report questionnaire) | Immediately after the intervention (3 weeks later)
  Coaches will complete acceptability measures via a self-report questionnaire, which will include close-ended questions rated on a scale of 1 (Strongly Disagree) to 5 (Strongly Agree; e.g., "The content was easy for athletes to understand and follow" and "The content covered topics that are important to my athletes") and open-ended questions (e.g., "What did you like about the Body Confident Athletes program and why?" and "What would you change about the Body Confident Athletes program and why?").
Total intervention fidelity (assessed via self-report and investigator observation of recorded intervention sessions) | Immediately after the intervention (3 weeks later)
  Total intervention fidelity will be assessed by the investigators through observing the program sessions as delivered by coaches and completing a pre-determined checklist to ensure the program was delivered to girls as intended. Additionally, girls will answer questions related to fidelity and comprehension (e.g., "Which Body Confident Athletes program sessions did you attend? Please select all that apply." and "In 2-3 sentences, what were the key topics discussed in the Body Confident Athletes program?").
Total intervention adherence (assessed through session completion) | Immediately after the intervention (3 weeks later)
  Total intervention adherence will be assessed by the investigators as the number of participants who complete the full intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Appearance Research, University of the West of England, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guthold R, Stevens GA, Riley LM, Bull FC. Global trends in insufficient physical activity among adolescents: a pooled analysis of 298 population-based surveys with 1.6 million participants. Lancet Child Adolesc Health. 2020 Jan;4(1):23-35. doi: 10.1016/S2352-4642(19)30323-2. Epub 2019 Nov 21. PMID 31761562
- [Background] Neumark-Sztainer D, MacLehose RF, Watts AW, Pacanowski CR, Eisenberg ME. Yoga and body image: Findings from a large population-based study of young adults. Body Image. 2018 Mar;24:69-75. doi: 10.1016/j.bodyim.2017.12.003. Epub 2017 Dec 27. PMID 29288970
- [Background] Sabiston, C., Pila, E., Vani, M., & Thogersen-Ntoumani, C. (2019). Body image, physical activity, and sport: A scoping review. Psychology Of Sport And Exercise, 42, 48-57. doi: 10.1016/j.psychsport.2018.12.010
- [Background] Sabiston, C. M., Vani, M. F., & Murray, R. M. (2021). Body-related self-conscious emotions in sport and exercise: A self-regulation perspective. In Motivation and Self-regulation in Sport and Exercise (pp. 62-77). Routledge.
- [Background] Slater A, Tiggemann M. Gender differences in adolescent sport participation, teasing, self-objectification and body image concerns. J Adolesc. 2011 Jun;34(3):455-63. doi: 10.1016/j.adolescence.2010.06.007. Epub 2010 Jul 31. PMID 20643477
- [Background] Vani MF, Pila E, Willson E, Sabiston CM. Body-related embarrassment: The overlooked self-conscious emotion. Body Image. 2020 Mar;32:14-23. doi: 10.1016/j.bodyim.2019.10.007. Epub 2019 Nov 13. PMID 31733410
- [Result] Matheson EL, Schneider J, Tinoco A, White P, Toher D, LaVoi NM, Diedrichs PC. A randomized controlled trial of a body image intervention for girl athletes. Health Psychol. 2025 Dec;44(12):1127-1138. doi: 10.1037/hea0001522. Epub 2025 Jun 2. PMID 40455543
- [Derived] Matheson EL, Schneider J, Tinoco A, Gentili C, Silva-Breen H, LaVoi NM, White P, Diedrichs PC. The co-creation, initial piloting, and protocol for a cluster randomised controlled trial of a coach-led positive body image intervention for girls in sport. BMC Public Health. 2023 Jul 31;23(1):1467. doi: 10.1186/s12889-023-16360-w. PMID 37525161